CLINICAL TRIAL: NCT00825877
Title: Long-Term Follow-Up of HALT-C Sustained Virologic Responders
Brief Title: Long-term Follow-up of HALT-C Sustained Virological Responders
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090067; 09-DK-0067
Record Dates: First submitted 2009-01-17; First posted 2009-01-21 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2012-06-29

CONDITIONS: Hepatitis C; Hepatocellular Carcinoma; Ascites; Variceal Hemorrhage; Death
Keywords: Hepatitis C; Sustained Virological Response; HALT-C; Peginterferon and Ribavirin; HCV RNA
MeSH Terms: conditions — Hepatitis C; Carcinoma, Hepatocellular; Ascites; Death

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
The Hepatitis C Antiviral Long-term Treatment against Cirrhosis (HALT-C) trial is a multicenter clinical trial conducted to assess the effects of long-term antiviral drug therapy on the progression of liver disease in patients who have advanced chronic hepatitis C and have not responded to prior therapies. Chronic hepatitis C is a long-lasting viral infection affecting the liver that may lead to permanent liver damage and cirrhosis (replacement of healthy liver cells by scar tissue). If left untreated, a proportion of patients with chronic hepatitis C will be at risk for complications of liver disease. The drug therapy in the HALT-C trial was designed to clear the hepatitis C virus from the patient s system in order to prevent or mitigate these potential complications. The purpose of this research is to determine if patients with chronic hepatitis C who experienced clearance of hepatitis C virus (known as a sustained virologic response, or SVR) during the HALT-C trial have developed any complications of their liver disease.

This study will include 180 subjects who participated in the initial phase of the HALT-C trial and experienced an SVR. The participants will visit the National Institutes of Health for an in-person study visit.

During the visit, patients will have blood drawn for lab tests to monitor the progress of their liver disease, and may be asked to undergo an ultrasound examination of the liver to detect any abnormalities that may be attributed to liver cancer. Patients will also answer questions about their medical history particularly any outcomes or events related to their hepatitis C that have occurred since the HALT-C trial and may be asked to sign a release of information to allow researchers to obtain medical records from other clinics or physicians where they have received treatment.

...

DETAILED DESCRIPTION:
Subjects who have achieved a sustained virologic response during their participation in the multicentered HALT-C clinical trial for treatment of chronic hepatitis C are being invited to return for a single clinic visit to assess whether any decompensation events (e.g. ascites, varicela hemorrhage, hepatic encephalopathy) or hepatocellular cancer has occurred. Subjects able and willing to return to the NIH will undergo standard clinical examinations, questionnaires and an ultrasound examination of the liver, to assess the status of their hepatitis C. Data will be pooled from all of the 10 clinical centers, analyzed and compared to an age and gender matched control group of nonresponder subjects who participated in the HALT-C Trial. A data coordinating center (New England Research Institutes) will conduct the data analysis. This will be a descriptive natural history study.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients who developed a virological response at week 20 of the HALT-C study.

EXCLUSION CRITERIA:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2009-01-15; Study Completion 2012-06-29

CONTACTS AND LOCATIONS:
Overall Officials: Marc G Ghany, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Morishima C, Morgan TR, Everhart JE, Wright EC, Shiffman ML, Everson GT, Lindsay KL, Lok AS, Bonkovsky HL, Di Bisceglie AM, Lee WM, Dienstag JL, Ghany MG, Gretch DR; HALT-C Trial Group. HCV RNA detection by TMA during the hepatitis C antiviral long-term treatment against cirrhosis (Halt-C) trial. Hepatology. 2006 Aug;44(2):360-7. doi: 10.1002/hep.21265. PMID 16871570
- [Background] Ikeda K, Saitoh S, Arase Y, Chayama K, Suzuki Y, Kobayashi M, Tsubota A, Nakamura I, Murashima N, Kumada H, Kawanishi M. Effect of interferon therapy on hepatocellular carcinogenesis in patients with chronic hepatitis type C: A long-term observation study of 1,643 patients using statistical bias correction with proportional hazard analysis. Hepatology. 1999 Apr;29(4):1124-30. doi: 10.1002/hep.510290439. PMID 10094956
- [Background] Yoshida H, Shiratori Y, Moriyama M, Arakawa Y, Ide T, Sata M, Inoue O, Yano M, Tanaka M, Fujiyama S, Nishiguchi S, Kuroki T, Imazeki F, Yokosuka O, Kinoyama S, Yamada G, Omata M. Interferon therapy reduces the risk for hepatocellular carcinoma: national surveillance program of cirrhotic and noncirrhotic patients with chronic hepatitis C in Japan. IHIT Study Group. Inhibition of Hepatocarcinogenesis by Interferon Therapy. Ann Intern Med. 1999 Aug 3;131(3):174-81. doi: 10.7326/0003-4819-131-3-199908030-00003. PMID 10428733